CLINICAL TRIAL: NCT00053131
Title: High Dose Cytarabine And Mitoxantrone Therapy For Relapsed And Refractory Acute Myeloid And Lymphocytic Leukemia: Effects Of GM-CSF Versus G-CSF On Dendritic Cells And Leukemia Associated Antigen-Specific T-Lymphocytes
Brief Title: Combination Chemotherapy Followed By Filgrastim or Sargramostim in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia or Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Maria Bear, MD, Roswell Park Cancer Institute
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000269285; RPCI-RPC-9902
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Filgrastim; sargramostim; Cytarabine; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Biological: sargramostim
Drug: cytarabine
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim and sargramostim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy. It is not yet known whether combination chemotherapy is more effective followed by filgrastim or sargramostim in treating leukemia.

PURPOSE: Randomized phase II trial to compare the effectiveness of combination chemotherapy followed by filgrastim with that of combination chemotherapy followed by sargramostim in treating patients who have relapsed or refractory acute myeloid leukemia or acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare amounts of dendritic cells and leukemia-associated antigen-specific T lymphocytes in patients with relapsed or refractory acute myeloid leukemia or acute lymphoblastic leukemia treated with filgrastim (G-CSF) vs sargramostim (GM-CSF) after high-dose cytarabine and mitoxantrone.

OUTLINE: This is a randomized study.

All patients receive high-dose cytarabine IV over 1 hour twice daily on days 1-6 and mitoxantrone IV over 30 minutes on days 2-4. On day 6, patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive filgrastim (G-CSF) subcutaneously (SC) daily until blood counts recover in the absence of unacceptable toxicity.
* Arm II: Patients receive sargramostim (GM-CSF) SC daily as in arm I.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia or acute lymphoblastic leukemia by morphology, cytochemical staining, and flow cytometry
* In first or subsequent relapse or refractory disease after at least 1 prior treatment regimen
* Antecedent hematologic disorders allowed except Philadelphia chromosome-positive chronic myelogenous leukemia

PATIENT CHARACTERISTICS:

Age

* 15 and over

Performance status

* 0-3

Life expectancy

* At least 4 weeks

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 2 times normal*
* SGOT no greater than 2 times normal* NOTE: *Unless directly attributable to leukemia

Renal

* Creatinine no greater than 1.5 times normal* NOTE: *Unless directly attributable to leukemia

Cardiovascular

* Ejection fraction at least 45%* NOTE: *Unless directly attributable to leukemia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent medical or psychiatric illness that would preclude study entry

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior autologous or allogeneic bone marrow or peripheral blood stem cell transplantation allowed
* Prior cytokines allowed

Chemotherapy

* Prior chemotherapy allowed

Endocrine therapy

* No concurrent corticosteroids except for treatment of severe vomiting that is refractory to standard agents

Radiotherapy

* Prior radiotherapy allowed

Surgery

* Not specified

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-01; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria R. Baer, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States